CLINICAL TRIAL: NCT00765908
Title: Ischaemic Pre-Conditioning in Elective PCI Patients - Attenuation of Subsequent Ischaemia in a Validated Animal Model
Brief Title: Ischaemic Pre-Conditioning in Elective Percutaneous Coronary Intervention (PCI) Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Dr Vladimir Dzavik, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UHN 2008-1
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients undergoing elective PCI will be randomised to 90 second balloon inflations rather than the standard less than 30 second inflations in order to induce peri-ischaemic conditioning.
  Interventions: Device: Angioplasty balloon
- B (Active Comparator): Control group. These patients will have a standard procedure with balloon inflations of 30 seconds or less as per standard.
  Interventions: Device: Angioplasty balloon

INTERVENTIONS:
Device: Angioplasty balloon — 90 second balloon inflation x 2
  Arms: A
Device: Angioplasty balloon — 30 seconds or less balloon inflations x 2
  Arms: B

SUMMARY:
This study aims to assess the potential for ischaemic peri-conditioning (IP) in elective percutaneous coronary intervention (PCI) patients to attenuate ischaemia in an animal model of myocardial infarct.

DETAILED DESCRIPTION:
Ischaemic preconditioning (IPC) was first described in a canine model by Murray et al in 1986. By deliberately inducing brief periods of myocardial ischaemia and reperfusion by intermittent occlusion of a coronary artery, the ability of the heart to withstand a subsequent, more prolonged episode of myocardial ischaemia was enhanced, to the extent that infarct size was reduced. This ubiquitous endogenous form of cardioprotection has been observed in many different species and is capable of limiting ischaemia-reperfusion in non-cardiac organs such as the brain, liver, gut, bladder and skin. It has been demonstrated to improve long term clinical outcomes in patients undergoing elective percutaneous coronary intervention (PCI)and to improve distal myocardial perfusion and mitigate infarct size in patients undergoing primary PCI . Despite extensive investigations into the cellular and molecular basis of IP, the precise mechanism(s) whereby myocytes develop tolerance to potentially fatal ischemia is unclear. There are also unanswered questions regarding the necessary frequency and duration of transient ischaemia needed to invoke the protection. Less than 60 seconds has been shown to be too short in some studies, whereas there is clearly an upper limit (above 10 minutes in most tissues) whereupon the preconditioning stimulus itself may have detrimental effects. Nonetheless, previous studies of IP in the heart have shown that a factor is released during IP, which can be transferred to protect another heart . Furthermore, preliminary data by our group suggests that 3 or 4 cycles of 5 minutes of transient limb ischaemia and 5 minutes of reperfusion (remote ischemic preconditioning, rIPC) leads to the release of a circulating cardioprotective factor(s) into the blood stream, which reduces cardiac damage in experimental animals, and patients undergoing cardiac surgery.

The proposed study will test whether these humoral factors are released from the heart, into the bloodstream, by patients undergoing PCI. The Langendorff method, in which a perfused rat heart is isolated ex vivo, is a well validated technique which has been used widely in studies of IP. It allows us to measure directly several cardiac physiological parameters, as well as the myocardial infarct size after prolonged ischaemia. We have previously shown that serum from healthy adults undergoing rIPC can be dialysed to produce a crystalloid perfusate. When this is used in the Langendorff preparation myocardial infarction size is reduced. We will employ the same method to examine the possible release, and any dose response to a pre-conditioning stimulus (coronary angioplasty balloon inflation) of varying duration in adults undergoing elective PCI.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent.
* All patients who are listed for elective PCI of at least one major epicardial artery.
* Patients ≥ 18 years and ≤80 years of age.

Exclusion Criteria:

* Any patient who has experienced chest pain within the preceding 24 hrs
* Any patient who exhibits haemodynamic instability (systolic BP <90mmHg, pulmonary oedema);
* Any patient with electrophysiologic instability (arrythmias eg rapid AF) or an abnormal baseline electrocardiogram (ECG) (e.g., significant ST segment depression, left bundle-branch block) which precludes analysis of the ST segment shift during PCI
* Patients unable to give informed consent
* Previous inclusion in this or any other clinical trial within one month prior to inclusion.
* Diabetes
* Uncontrolled hypertension (BP>180/110).
* Anaemia (Hb <10g/l).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Attenuation of infarct size and improved post-ischemia haemodynamic recovery in rat hearts. | immediate

SECONDARY OUTCOMES:
Clinical endpoints: (i) induction of IP, defined as a minimum 33% reduction in magnitude of ST segment deviation in the territory of the affected artery between the first and second balloon inflation. (ii) Reduction in CK rise post procedure. | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dzavik, MD, Principal Investigator — University Health Network, Toronto